CLINICAL TRIAL: NCT00481143
Title: A One-year, Open-label, Single Arm, Multi-center Trial Evaluating the Efficacy and Safety of Oral ICL670 in Patients Diagnosed With Low and INT-1 Risk Myelodysplastic Syndrome (MDS) and Transfusion-dependent Iron Overload
Brief Title: Efficacy and Safety of Deferasirox in Patients With Myelodysplastic Syndrome and Transfusion-dependent Iron Overload
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ADE03
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2016-11

CONDITIONS: Myelodysplastic Syndromes; Transfusion Dependent Iron Overload
Keywords: Myelodysplastic Syndrome; MDS; iron overload; chelation; chelators; ICL670; Deferasirox; serum ferritin; LIC; transfusional hemosiderosis; Refractory Anemia; RA; Refractory Anemia with Ringed Sideroblasts; RARS; blood transfusions; Mydelodysplastic Syndrome(s)
MeSH Terms: conditions — Myelodysplastic Syndromes; Iron Overload; Anemia, Refractory | interventions — Deferasirox

ARMS (1):
- deferasirox (Experimental)
  Interventions: Drug: ICL670/Deferasirox

INTERVENTIONS:
Drug: ICL670/Deferasirox
  Other Names: ICL670

SUMMARY:
The purpose of this study is to investigate the effects of iron chelation using deferasirox in low and INT-1 risk (referring to the international prognostic scoring system, IPSS) MDS patients who show signs of iron overload due to repeated blood transfusions.

This trial is not recruiting patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

* MDS patients presenting with low or intermediate-1 IPSS risk and transfusional iron overload
* Patients of either gender and age ≥ 18 years
* History of at least 20 units of red blood cell transfusions or 100mL/kg of prepacked red blood cells (PRBCs)
* Patients can be either naïve to iron chelation or have had prior treatment with deferoxamine (DFO) or deferiprone (L1)
* Females of childbearing potential must use double-barrier contraception, oral contraceptive plus barrier contraceptive, or must have undergone clinically documented total hysterectomy and/or oophorectomy, tubal ligation or be postmenopausal defined by amenorrhea for at least 12 months.

Exclusion Criteria:

* Non-transfusion related iron overload
* Treatment with deferasirox (ICL670) before study start
* Patients with a concomitant malignant disease
* Patients with out of range lab values
* History of nephrotic syndrome
* Patients with a previous history of clinically relevant ocular toxicity related to iron chelation
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent the patient from undergoing study treatment
* Patients treated with systemic investigational drugs within the past 4 weeks or topical investigational drug within the past 7 days
* Any other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug.
* Patients with active uncontrolled infectious disease
* Pregnancy or breast feeding

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To assess iron chelation by comparing serum ferritin values at baseline vs. 52 weeks of treatment with deferasirox | 52 weeks

SECONDARY OUTCOMES:
Safety and tolerability of deferasirox assessed by monitoring and recording all adverse events (AEs) and serious adverse events (SAEs) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany

REFERENCES:
- [Result] Nolte F, Hochsmann B, Giagounidis A, Lubbert M, Platzbecker U, Haase D, Luck A, Gattermann N, Taupitz M, Baier M, Leismann O, Junkes A, Schumann C, Hofmann WK, Schrezenmeier H. Results from a 1-year, open-label, single arm, multi-center trial evaluating the efficacy and safety of oral Deferasirox in patients diagnosed with low and int-1 risk myelodysplastic syndrome (MDS) and transfusion-dependent iron overload. Ann Hematol. 2013 Jan;92(2):191-8. doi: 10.1007/s00277-012-1594-z. Epub 2012 Oct 17. PMID 23073603